CLINICAL TRIAL: NCT05589584
Title: Effect of N-acetyl Cysteine on Markers of Oxidative Stress and Insulin Resistance in Patients with Non-alcoholic Fatty Liver Disease
Brief Title: N-acetyl Cysteine and Patients with Non-alcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Asmaa Mohammad Ramadan, hospital pharmacist, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1234867
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2022-10

CONDITIONS: Simple Steatosis Non Fatty Liver
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention (Experimental): NAC and weight reduction program
  Interventions: Drug: N acetyl cysteine with weight reduction
- control (No Intervention): weight reduction program only

INTERVENTIONS:
Drug: N acetyl cysteine with weight reduction — high dose 2400mg/day
  Arms: intervention

SUMMARY:
Effect of N-acetyl cysteine on markers of oxidative stress and insulin resistance in patients with Non-alcoholic fatty liver disease

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18-60 years diagnosed with NAFLD

Exclusion Criteria:

* History of alcohol consumption, drug addiction or the use of medications known to precipitate steatohepatitis.
* Patients with schistosomiasis, active hepatitis B or C, autoimmune and diabetes mellitus.
* current Consumption of any antioxidant supplements and hepatotoxic drug.
* Pregnancy or lactation or expecting to get pregnant during the study.
* Medical, psychological, or pharmacological factors interfering with the collection or interpretation of study data.
* Active Cancer patients.
* Anyone having hypersensitivity to N-acetylcysteine.
* Anyone already taking N-acetylcysteine.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
assessment of the effect of NAC on leptin | 3 months
  leptin as insulin resistance marker in NAFLD

SECONDARY OUTCOMES:
assessment of the effect of NAC on MDA | 3 months
  MDA as oxidative stress marker in NAFLD

CONTACTS AND LOCATIONS:
Locations (1):
- NHTMRI, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No